CLINICAL TRIAL: NCT05848895
Title: OPT-IN: Osteopathic Plagiocephaly Treatment for Infants and Neonates
Acronym: OPT-IN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Osteopathy's Promise to Children (Other)
Responsible Party: Principal Investigator, Kimberly Wolf, Kimberly Wolf, DO, Osteopathy's Promise to Children
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: OPC001
Record Dates: First submitted 2023-04-28; First posted 2023-05-08 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-03

CONDITIONS: Plagiocephaly, Nonsynostotic; Plagiocephaly, Positional; Plagiocephaly; Cranium; Deformity
Keywords: Positional Plagiocephaly; Nonsynostotic Plagiocephaly; Repositioning; Osteopathic Manipulative Treatment; Cranial asymetry
MeSH Terms: conditions — Plagiocephaly, Nonsynostotic; Plagiocephaly; Congenital Abnormalities | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Osteopathic Manipulative Treatment (Experimental): Patients will be treated once a week with OMT x 8 weeks
  Interventions: Procedure: Osteopathic Manipulative Treatment
- Standard of Care Repositioning (Active Comparator): Patients will only receive repositioning only x 8 weeks and all parents will receive standardized materials to counsel/instruct on the repositioning
  Interventions: Behavioral: Standard of Care Repositioning

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment — Osteopathic Manipulative Treatment is a manual treatment therapy applied by licensed physicians that consists of using ones hands to improve the structure and function of the body. In this situation it will involve gentle and passive modalities that are well-tolerated by infants.
  Arms: Osteopathic Manipulative Treatment
Behavioral: Standard of Care Repositioning — Parents will receive standardized handouts/materials instructing on repositioning intended to help improve head shape in infants with plagiocephaly.
  Arms: Standard of Care Repositioning

SUMMARY:
The goal of this crossover randomized clinical trial is to assess the effects of osteopathic manipulative treatment (OMT) compared to standard of care repositioning in children diagnosed with positional/deformational plagiocephaly. The main hypothesis is that children who received OMT will show significantly improved anthropometric measures of cranial symmetry over those receiving the current pediatric standard of care of repositioning.

This is a two-arm, randomized cross-over clinical trial. With parental consent, pediatric patients (infants <4 months of age) will be organized into one of two groups:

1. Those who receive OMT with emphasis on osteopathic cranial manipulative medicine (OCMM) to restore cranial symmetry.
2. Those who receive standard care only with repositioning attention from the parents After 8-weeks of being in the first group, each participant will cross-over into the second group (OMT or repositioning) N = 122 subjects diagnosed with deformational plagiocephaly (DP) are to be recruited (to allow for natural attrition and loss to follow up) with the recruitment to continue until 61 patients have been placed in each of the two groups and will cross-over to the respective treatment group (OMT and standard of care repositioning therapy).

Timeline: It is projected that to recruit and carry out the assessments and interventions (8-weeks of each group with 12-months of follow-up longitudinally), it will require two years (24-months) from the beginning of the study to completion.

ELIGIBILITY:
Inclusions:

* Diagnosed with positional plagiocephaly
* Under 4-months of age (between birth - 4 months) at the time of enrollment

Exclusions:

* Preterm birth (<37 weeks)
* Genetic syndromes
* Craniofacial defects/deformities (e.g. cleft lip/palate)
* Brachycephaly/scaphocephaly
* Hypotonia
* Hypertonia
* Craniosynostosis
* Head trauma or other neurological illnesses
* Lost to follow up
* Patient whose parents (or legal guardians) disagree to attend 8-treatments of OMT and 2 additional measurement sessions
* Prior helmet therapy, physical therapy, or OMT before the date of enrollment

Ages: 1 Day to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 122 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cranial Vault Asymmetry Index | 2 years
  Anthropometric measurement of cranial asymmetry
Head circumference | 2 years
  Standard growth parameter measured in infants
Weight | 2 years
  Standard growth parameter measured in infants

SECONDARY OUTCOMES:
Medical history | 12 months
  Patients charts will be reviewed after first year of life to assess for medical issues including otitis media, developmental delay, allergic rhinitis, vision problems, torticollis, hospitalizations, need for a helmet to treat plagiocephaly, colic, reflux/GER, etc.
Developmental Milestones | 12 months
  Patients' enrolled in the study will have developmental stones monitored as per general pediatrician's protocol to screen for developmental delays.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly J Wolf, DO, Principal Investigator — Osteopathy's Promise to Children
Locations (1):
- Osteopathic Center San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No